CLINICAL TRIAL: NCT00515125
Title: A Randomised Trial of Oral Nutritional Supplements Versus Dietary Advice on Clinical Nutrition in the Community.
Brief Title: Community Oral Nutrition Support Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELIA0001
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-06

CONDITIONS: Malnutrition
Keywords: Quality of life; Supplement; Care home; Elderly; Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Nutrition Assessment; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Advice (Other): Dietary Advice
  Interventions: Behavioral: Dietary Advice
- Oral Nutritional Supplements (Other): Oral Nutritional Supplements
  Interventions: Dietary Supplement: Oral Nutritional Supplements (Fortisip)

INTERVENTIONS:
Behavioral: Dietary Advice — Dietary Advice sheet
  Arms: Dietary Advice
Dietary Supplement: Oral Nutritional Supplements (Fortisip) — These products are classified as non-medicinal, borderline substances, foods for special medical purposes.
  A range of commercially available liquid oral nutritional supplements (Fortisip) will be offered daily for a 12 week period.
  Arms: Oral Nutritional Supplements

SUMMARY:
The purpose of this study is to determine the best form of dietary intervention to undernourished elderly individuals in care homes.

The research aims to test the null hypothesis that there is no difference between oral nutritional supplements and dietary advice as the first line treatment for malnutrition.

DETAILED DESCRIPTION:
A prospective, randomised, parallel, open-label trial, study in malnourished care home residents, without obvious dementia, to compare the effects of two common forms of nutritional support; dietary advice (DA) and oral nutritional supplements (ONS), on quality of life (QoL) and other outcomes including weight, nutritional intake and appetite. The residents were randomised to receive either DA provided by a dietitian or ONS for a period of 12 weeks. The primary outcome measure was QoL and the secondary outcome measure was dietary intake.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age > 50 years
* At risk of malnutrition
* Competent to provide written informed consent and to answer questions
* Able to eat and drink
* Willingness to take part in the trial and to follow the trial protocol

Exclusion Criteria:

* Requirement for tube or parenteral nutrition
* Galactosemia
* Receiving current oral nutritional supplementation
* Palliative care
* Chronic renal disease requiring dialysis
* Liver failure
* Malignancy
* Participation in other studies

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is Quality of Life | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marinos Elia, Professor, Principal Investigator — University of Southampton
Locations (1):
- Care Homes in Hampshire, Southampton, Hampshire, United Kingdom

REFERENCES:
- [Derived] Parsons EL, Stratton RJ, Cawood AL, Smith TR, Elia M. Oral nutritional supplements in a randomised trial are more effective than dietary advice at improving quality of life in malnourished care home residents. Clin Nutr. 2017 Feb;36(1):134-142. doi: 10.1016/j.clnu.2016.01.002. Epub 2016 Jan 11. PMID 26847947